CLINICAL TRIAL: NCT03574116
Title: Could a Preoperative Feeding Jejunostomy Decrease Sarcopenia for Patients With Oesogastric Adenocarcinoma ?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6808
Record Dates: First submitted 2018-05-31; First posted 2018-06-29 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-05

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; jejunostomy; oesogastric adenocarcinoma; scanography
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study of sarcopenia is a subject that is the subject of numerous research and publications, particularly because of its link with a poor prognosis for many cancers.

In an article published by the digestive surgery team, the role of feeding jejunostomy has been demonstrated: it allowed more patients to reach the 2nd stage of surgery and a better tolerance of chemotherapy.

Investigators wanted to study retrospectively the impact of feeding jejunostomy on radiological sarcopenia. Is the positive effect of jejunostomy in gastric cancers associated with a decrease in sarcopenia?

ELIGIBILITY:
Criteria for inclusion:

* Age 18-80 years
* Sex: H or F
* Subject giving their consent for their participation
* Gastric cancers
* stage> IB
* whether or not a feeding jejunostomy
* CT scan performed at the HUS, after the end of the courses of chemotherapy and / or before the surgery.

Exclusion criteria:

* antecedent level L3 surgery,
* psoas hematoma
* No CT performed at HUS at the end of chemotherapy and / or before surgery
* Impossibility of giving the subject informed information
* Subject under the protection of justice
* Subject under guardianship or curatorship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with Stage IB Gastric Cancer and having benefited from the placement or not of a feeding jejunostomy and a control CT performed at the HUS, after the end of the courses of chemotherapy and / or before the surger
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate muscle status by CT evaluation of sarcopenia in patients | 24 hour after the realization of the MRI
  Evaluate the impact of feeding jejunostomy in patients with gastric cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Service Imagerie 1, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No